CLINICAL TRIAL: NCT05411393
Title: Synergizing Home Health Rehabilitation Therapy to Optimize Patients' Activities of Daily Living
Brief Title: Synergizing Home Health Rehabilitation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202102816 -N; R21AG076972 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Frailty; Frail Elderly; Occupational Therapy; Activities of Daily Living; Home Health Care; Functional Status; Physical Functional Performance; Rehabilitation; Treatment Outcome; Health Services for the Aged
Keywords: Rehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Experimental arm versus the control arm
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the group allocation of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Research participants in this arm will receive the ADL-enhanced program and usual home health care rehabilitation. The ADL-enhanced program consists of six home visits delivered by a study occupational therapist.
  Interventions: Other: ADL-enhanced program; Other: Usual home health rehabilitation therapy
- Control arm (Other): Research participants in this arm will receive usual home health care rehabilitation.
  Interventions: Other: Usual home health rehabilitation therapy

INTERVENTIONS:
Other: ADL-enhanced program — The ADL-enhanced program consists of six home visits delivered by a study occupational therapy staff. The study therapy staff will use the compensatory approach and the restorative approach during the visits to enhance patients' activity engagement. The compensatory approach uses strategies to reduce the activity demand to make every task easier. For example, using the sitting position to perform self-care tasks. The restorative approach uses strategies to increase the demand of the task to increase the patient's functional capacity. For example, carrying a full-load laundry basket versus an empty laundry basket.
  Arms: Experimental arm
Other: Usual home health rehabilitation therapy — Usual home health rehabilitation therapy is prescribed by the home health agency. It often includes occupational therapy and physical therapy delivered in one to three home visits per week for one to two months.

SUMMARY:
The objective of this project is to pilot test an ADL (activities of daily living)-enhanced program as an adjuvant therapy to usual home health rehabilitation to improve patient outcomes. The project will compare the ADL-enhanced program plus usual care with usual care using an RCT design in home health patients.

DETAILED DESCRIPTION:
Regaining the ability to take care of oneself after an illness or medical episode is critical for home health patients to maintain independent living at home. An ADL-enhanced program may augment the effect of home health rehabilitation therapy to support patients' self-care outcomes. Patients will be randomly assigned to two groups: one will receive the ADL-enhanced program with usual home health care, and the other will receive usual home health care. Researchers will compare outcomes in self-care activities and physical performance between the two groups to determine the effect of the ADL-enhanced program.

ELIGIBILITY:
Patients are eligible if they

* are 65 years of age over older
* are Medicare beneficiaries
* are referred for skilled rehabilitation services at the partnered home health agency
* have three or more comorbidities

Patients are ineligible if they have

* acute fractures with surgical or weight-bearing restrictions,
* elective joint replacement surgery
* lower-extremity amputation
* active treatment for cancer diagnosis
* ongoing dialysis treatment
* acute cardiac surgery,
* acute stroke or a major neurologic disorder limiting motor movements
* terminal stage of congestive heart failure
* a referral to hospice care
* severe cognitive deficits limiting verbal communication.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-ju Liu, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 6, 2022, and October 15, 2024, 47 Medicare patients were recruited from partnered home health agencies.
Pre-assignment Details: There is no pre-assignment. After baseline assessment, participants were randomly assigned to the experimental group or the control group.
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started | 24 | 23
Completed | 18 | 21
Not Completed | 6 | 2
Not completed — Illness or loss of interest | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental Arm: Research participants in this arm received the ADL-enhanced program and usual home health care rehabilitation. The ADL-enhanced program consists of six home visits delivered by a study therapy interventionist.
  ADL-enhanced program: The ADL-enhanced program consists of six home visits delivered by a study therapy staff. The study therapy staff used the compensatory approach and the restorative approach during these visits to enhance patients' activity engagement. The compensatory approach includes strategies to reduce the activity demand to make every task easier. For example, using the sitting position to perform self-care tasks. The restorative approach uses strategies to increase the demand of the task to increase the patient's functional capacity. For example, carrying a full-load laundry basket versus an empty laundry basket.
  Usual home health rehabilitation therapy: Usual home health rehabilitation therapy was prescribed by the home health agency. It often included occupational therapy and physical therapy delivered in one to three home visits per week for one to two months.
- Control Arm: Research participants in this arm received usual home health care rehabilitation.
  Usual home health rehabilitation therapy: Usual home health rehabilitation therapy was prescribed by the home health agency. It often included occupational therapy and physical therapy delivered in one to three home visits per week for one to two months.
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.6 (8.2) | 83.1 (6.9) | 82.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 16 | 19 | 35
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 0 | 0 | 0
Years of education [Mean (Standard Deviation); unit: Years] | 14.6 (3.4) | 15.2 (2.7) | 14.9 (3.1)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per square meter] | 26.7 (5.8) | 25.5 (5.6) | 26.1 (5.7)
Number of self-reported chronic conditions [Mean (Standard Deviation); unit: The number of chronic conditions] | 5.3 (2.2) | 5.6 (2.5) | 5.4 (2.3)
The number of medications currently taken [Mean (Standard Deviation); unit: The number of medications] | 8 (3.9) | 8.3 (4.5) | 8.2 (4.1)
Pain, Enjoyment of Life, and General Activity Scale [Mean (Standard Deviation); unit: Score on the scale] — A pain scale with a possible score ranging from 0 to 10. A higher score indicates a higher degree of pain.
  Score on the scale | 4 (3.1) | 3.6 (3.2) | 3.8 (3.1)
The Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: Score] — A depression measure with a possible score ranging from 0 to 27. A higher score indicates a higher degree of depression.
  Score | 6.4 (5.2) | 7.1 (5.5) | 6.7 (5.3)
Saint Louis University Mental Status Exam [Mean (Standard Deviation); unit: Score] — A global cognition measure with a possible score ranging from 0 to 30. A higher score indicates better cognitive function.
  Score | 21.9 (6.1) | 22.9 (5) | 22.4 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: The Motor Skills Score From the Assessment of Motor and Process Skills
Description: The Motor Skills score is a subscale in the Assessment of Motor and Process Skills, which evaluates the degree of motor performance when an individual performs a challenging daily activity. The score range of the subscale ranges from -3 to +4. A higher score indicates better motor performance.
Time Frame: Baseline, post-intervention (approximately 2 months from baseline), and 1-month follow-up (approximately 3 months from baseline)
Population: At post-intervention assessments, three participants in the treatment group did not complete the assessment. At 1-month follow-up, five participants in the treatment group and one in the control group did not complete the assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
Units on a scale
  Baseline | 1.3 (0.4) | 1.1 (0.5)
  Post-intervention: number analyzed (Participants) | 21 | 23
  Post-intervention | 1.3 (0.5) | 1.4 (0.5)
  1-month follow up: number analyzed (Participants) | 19 | 22
  1-month follow up | 1.5 (0.5) | 1.5 (0.6)

2. Secondary Outcome: Activity Measure Post Acute Care: Home Care Short Form
Description: Activity Measure Post Acute Care: Home Care Short Form is a self-reported outcome measure of functional independence to live in the community. The reported T-score is a standardized score derived from raw responses, scaled to have a mean of 50 and a standard deviation of 10 in the reference population. The Basic Mobility subscale evaluates indoor and outdoor mobility; higher scores indicate better mobility performance. The Daily Activity subscale measures the ability to perform self-care tasks at home; higher scores reflect better performance in daily activities.
Time Frame: Baseline, post-intervention (approximately 2 months from baseline), 1-month follow-up (approximately 3 months from baseline), 3-month follow-up (approximately 5 months from baseline)
Population: At post-intervention assessments, three participants in the treatment group did not complete the assessment. At 1-month follow-up, five participants in the treatment group and one in the control group did not complete the assessment. At 3-month follow-up, six participants in the treatment group and two in the control group did not complete the assessment.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
T Score
  Basic mobility subscale at baseline | 51.2 (7.0) | 49.5 (6.6)
  Basic mobility subscale at post-intervention: number analyzed (Participants) | 21 | 23
  Basic mobility subscale at post-intervention | 51.8 (5.7) | 52.2 (8.0)
  Basic mobility subscale at 1-month follow-up: number analyzed (Participants) | 19 | 22
  Basic mobility subscale at 1-month follow-up | 52.0 (4.3) | 52.5 (9.0)
  Basic mobility subscale at 3-month follow-up: number analyzed (Participants) | 18 | 21
  Basic mobility subscale at 3-month follow-up | 54.2 (6.4) | 54.8 (8.2)
  Daily activity subscale at baseline | 48.7 (8.0) | 47.5 (8.9)
  Daily activity subscale at post-intervention: number analyzed (Participants) | 21 | 23
  Daily activity subscale at post-intervention | 51.1 (7.7) | 50.6 (8.7)
  Daily activity subscale at 1-month follow-up: number analyzed (Participants) | 19 | 22
  Daily activity subscale at 1-month follow-up | 51.2 (8.5) | 51.1 (8.7)
  Daily activity subscale at 3-month follow-up: number analyzed (Participants) | 18 | 21
  Daily activity subscale at 3-month follow-up | 49.1 (8.6) | 52.7 (8.8)

3. Secondary Outcome: Box and Block Test
Description: The test measures motor coordination of the upper extremity through moving small wooden blocks within one minute. Each hand was tested separately. A higher score indicates better hand function.
Time Frame: as for outcome 1
Population: The data reported here are based on participants who were able to complete the test at each time point.
Measure: Mean (Standard Deviation); unit: The number of blocks
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
The number of blocks
  Right hand at baseline: number analyzed (Participants) | 23 | 23
  Right hand at baseline | 40.1 (7.2) | 38.6 (9.5)
  Right hand at post-intervention: number analyzed (Participants) | 20 | 23
  Right hand at post-intervention | 41.9 (8.7) | 39.5 (7.4)
  Right hand at 1-month follow-up: number analyzed (Participants) | 19 | 21
  Right hand at 1-month follow-up | 41.3 (7.9) | 39.15 (9.2)
  Left hand at baseline: number analyzed (Participants) | 23 | 23
  Left hand at baseline | 39.6 (7.0) | 36.3 (9.1)
  Left-hand at post-intervention: number analyzed (Participants) | 20 | 23
  Left-hand at post-intervention | 39 (8.9) | 36.8 (9.1)
  Left-hand at 1-month follow-up: number analyzed (Participants) | 19 | 21
  Left-hand at 1-month follow-up | 36.8 (11.6) | 38.3 (9.0)

4. Secondary Outcome: Jebsen Hand Function Test
Description: The test measures upper extremity function by recording the time it takes to complete seven daily tasks, such as writing or picking up small, common objects. A longer time to complete all tasks indicates poor hand function.
Time Frame: as for outcome 1
Population: The data reported here are based on participants who were able to complete the test at each time point.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
Seconds
  Baseline | 82.7 (49.7) | 84.0 (25.0)
  Post-intervention: number analyzed (Participants) | 21 | 23
  Post-intervention | 86.9 (60.0) | 83.0 (28.6)
  1-month follow-up: number analyzed (Participants) | 19 | 21
  1-month follow-up | 88.9 (72.6) | 78.0 (22.8)

5. Secondary Outcome: Timed-Up-and-Go Test
Description: The test measures functional mobility by recording the time it takes to get up from a chair, walk, and return to the chair. A higher score indicates poor functional mobility.
Time Frame: as for outcome 1
Population: The data reported here are based on participants who were able to complete the test at each time point.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
Seconds
  Baseline: number analyzed (Participants) | 23 | 22
  Baseline | 24.5 (13.2) | 30.6 (18.7)
  Post-intervention: number analyzed (Participants) | 20 | 22
  Post-intervention | 22.8 (9.3) | 24.7 (13.4)
  1-month follow-up: number analyzed (Participants) | 19 | 20
  1-month follow-up | 24.2 (10.9) | 23.5 (14.4)

6. Secondary Outcome: Short Physical Performance Battery
Description: The test measures balance, walking speed and chair stand. The score range is from 0 to 12. A higher score indicates better physical performance of the lower extremity.
Time Frame: as for outcome 1
Population: The data reported here are based on participants who were able to complete the test at each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 24 | 23
Score on a scale
  Baseline | 3.7 (2.2) | 4.0 (2.5)
  Post-intervention: number analyzed (Participants) | 21 | 23
  Post-intervention | 4.1 (1.7) | 4.6 (2.6)
  1-month follow up: number analyzed (Participants) | 19 | 21
  1-month follow up | 4.3 (1.9) | 4.9 (2.8)

ADVERSE EVENTS:
Time Frame: From baseline until 3-month follow-up, about 5 months.
Arm/Group | Experimental Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT05411393/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT05411393/ICF_000.pdf